CLINICAL TRIAL: NCT03899740
Title: OCS-Tapering-Delphi: Expert Statements Concerning the Tapering of Oral Corticosteroids (OCS) for the Treatment of Asthma: A Delphi Consensus Study
Brief Title: Expert Statements Concerning the Tapering of Oral Corticosteroids (OCS) for the Treatment of Asthma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association Jean Baptiste Desbrest (Other)
Collaborators: AstraZeneca (Industry); University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: JDB-Delphi-201903
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The expert panel: Participation in this study will be proposed to a group of experts, including pulmonologists, endocrinologists, allergists, paediatricians and rheumatologists. Additionally, patient advocacy organization representatives will also be invited.
  Experts meeting eligibility criteria (see section below) are invited to participate. Further details are available via the URL link at the end of this declaration.
  Interventions: Other: Brainstorming 1; Other: Ranking - Round 1; Other: Ranking - Round 2; Other: Ranking - Round 3

INTERVENTIONS:
Other: Brainstorming 1 — Expert recommendation statements will be collected for peer evaluation.
Other: Ranking - Round 1 — Each participant will rank each statement using a likert scale: strongly disagree -- disagree -- neutral -- agree -- strongly agree.
Other: Ranking - Round 2 — Each participant will rank each statement using a likert scale: strongly disagree -- disagree -- neutral -- agree -- strongly agree.
Other: Ranking - Round 3 — Each participant will rank each statement using a likert scale: strongly disagree -- disagree -- neutral -- agree -- strongly agree.

SUMMARY:
The objectives of this study are to use the Delphi method to assemble an expert panel representing innovation in asthma treatment, to collect freely suggested recommendation statements concerning OCS tapering (and sub-topics) among severe asthma patients from this panel for peer evaluation, and finally to determine the level of consensus for each statement from the panel as a whole.

DETAILED DESCRIPTION:
A series of anonymous questionnaires will be administered to a panel of experts. Each questionnaire administered results in a body of information that is re-presented to the experts before performing the next round. Initial brainstorming questionnaires are open in nature, and are used to generate statements that individual experts would like to see evaluated by their peers. Subsequent ranking questionnaires require that each expert rank each statement according to a pre-defined likert scale. Serial ranking questionnaires are administered electronically and continue until stopping rules are met, or the maximum number of allowed rounds is achieved (capped at three rounds for the present study).

Experts are recruited by invitation or response to open call (see eligibility criteria and url at the end of this declaration.)

ELIGIBILITY:
Inclusion Criteria:

* The expert is either a pulmonologist/respiratory disease specialist, an allergist, an endocrinologist, a paediatrician, a rheumatologist or a patient advocacy organisation representative
* All clinicians involved must manage patients on a weekly basis and have clinical experience in managing disease following oral corticosteroid withdrawal/tapering.
* Patient advocacy organization representatives must represent a relevant patient group (and provide contact information for their group)

Exclusion Criteria:

* Currently employed by a pharmaceutical company, or will have such employment in the upcoming 12 months
* Ownership in a pharmaceutical company or any other conflict of interest with the present study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The expert panel may include pulmonologists, endocrinologists, allergists, paediatricians and rheumatologists. Additionally, patient advocacy organization representatives will also be invited.
  Potential experts may respond to open invitation via the link at the end of this study registration.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-09-26 (Estimated); Study Completion 2019-09-26 (Estimated)

PRIMARY OUTCOMES:
The number of recommendation statements achieving positive consensus | Approximately month 5
  When >= 70% of the expert panel indicates either "agree" or "strongly agree" for a given statement, a positive consensus has been met.
The number of recommendation statements achieving negative consensus | Approximately month 5
  When >= 70% of the expert panel indicates either "disagree" or "strongly disagree" for a given statement, a positive consensus has been met.
The number of recommendation statements achieving consensus for neutrality | Approximately month 5
  When >= 70% of the expert panel indicates "neutral" for a given statement, a consensus for neutrality has been met.

SECONDARY OUTCOMES:
The number of statements meeting the stopping rule after ranking round 1. | Approximately month 5
  When >= 70% of the expert panel indicates the same score for a given statement, no subsequent rounds of ranking for that statement will be performed.
The number of statements meeting the stopping rule after ranking round 2. | Approximately month 5
  When >= 70% of the expert panel indicates the same score for a given statement, no subsequent rounds of ranking for that statement will be performed.
The number of statements meeting the stopping rule after ranking round 3. | Approximately month 5
  When >= 70% of the expert panel indicates the same score for a given statement, no subsequent rounds of ranking for that statement will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carey Suehs, PhD, Study Director — Association Jean Baptiste Desbrest
Locations (1):
- Association Jean Baptiste Desbrest, Montpellier, France

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on an appropriate public platform at the time of publication.
Supporting Information: Study Protocol
Time Frame: Anonymized data will be shared on an appropriate public platform at the time of publication.
URL: https://osf.io/wrdbu/

REFERENCES:
- See also: The OCS Tapering Delphi study on the Open Science Framework. — https://osf.io/wrdbu/